CLINICAL TRIAL: NCT05636696
Title: COMPANION Study: A Pilot Trial Testing Couple Mindfulness-based Cognitive Behavioral Therapy Via Internet Targeting Cancer-related Fatigue [Workpackage 2]
Brief Title: COMPANION: A Couple Intervention Targeting Cancer-related Fatigue
Acronym: COMPANION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mariët Hagedoorn (Other)
Collaborators: Helen Dowling Institute (Unknown)
Responsible Party: Sponsor-Investigator, Mariët Hagedoorn, Principal Investigator, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202100817; KWF-12794 (Other Grant/Funding Number: Dutch Cancer Society); NL80201.042.22 (Other: CCMO register (ABR))
Record Dates: First submitted 2022-10-31; First posted 2022-12-05 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Neoplasms; Fatigue
Keywords: Chronic cancer-related fatigue; Cancer; Behavioral intervention; Mindfulness intervention; Dyadic intervention; Pilot; Partners; Spouses
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Intervention Model Description: This is a 1-arm pilot trial. All eligible and consenting couples will be allocated to the couple eMBCT named 'COMPANION' (Dutch name: 'Samen Minder Moe'). No randomization takes place.
  The couple eMBCT was developed based on the evidence-based eMBCT directed (only) at patients. The couple eMBCT entails nine sessions, takes 15-20 weeks, can be followed from home and will be supervised remotely by a trained psychotherapist. Consistent with the original (patient only) eMBCT, the couple eMBCT aims to change the patient's behavioral and cognitive reactions to fatigue and other cancer-related stressors. Couple eMBCT includes extra information for partners each session, the possibility for partners to perform exercises and one extra session dedicated to the couple's mutual relationship and mindful communication about CCRF. Couples can determine themselves to which degree the partner is involved in the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- couple eMBCT (Experimental): The couple eMBCT has nine sessions, takes 15-20 weeks, can be followed from home and will be supervised remotely by a trained therapist. Consistent with the original (patient-only) eMBCT, the couple eMBCT aims to change the patient's behavioral and cognitive reactions to fatigue and other cancer-related stressors. Couple eMBCT includes information for partners each session, the possibility for partners to perform exercises and one session specifically dedicated to the couple's mutual relationship and mindful communication about CCRF. Couples can determine themselves to which degree the partner is involved in the therapy.
  Interventions: Behavioral: Samen Minder Moe (Dutch intervention name)

INTERVENTIONS:
Behavioral: Samen Minder Moe (Dutch intervention name) — 'Samen Minder Moe' is a mindfulness-based cognitive behavioral therapy for cancer-related fatigue directed at couples.
  Other Names: COMPANION; couple eMBCT

SUMMARY:
Chronic cancer-related fatigue (CCRF) is a disturbing condition that persists in up to 25% of cancer patients after completion of treatment. While mindfulness-based interventions are effective in relieving CCRF, these typically target the patient alone. Growing evidence suggests that including partners and targeting the dyadic context can increase and broaden the interventions' efficacy. The proposed study is a pilot trial testing the acceptability and potential efficacy of a mindfulness intervention directed at couples.

DETAILED DESCRIPTION:
This is a 1-arm pilot trial. Recruitment will take place via a hospital, the Helen Dowling Institute and self-referral. The target is to include 34 couples (i.e. 68 participants). All participating cancer patients and their partners will be allocated to the couple mindfulness-based cognitive behavioral therapy, provided via internet (couple eMBCT), called 'COMPANION' (in Dutch: 'Samen Minder Moe') Assessments include three questionnaires (i.e. before starting the intervention (T0), after completing the intervention (T1), and 1 month after T1 (T2)). The assessments include also weekly diaries during a period of 17-22 weeks. A subsample of patients (n ≈ 5) and partners (n ≈ 5) as well as the therapists providing the couple eMBCT will participate in final focus groups. The primary objectives of COMPANION study 2 are to determine the acceptability of the couple intervention and the potential efficacy for patient fatigue. Secondary objectives are to examine the feasibility of trial procedures and the potential working mechanisms of the couple intervention.

ELIGIBILITY:
Inclusion Criteria:

Only couples are eligible for participation. In order to be eligible, the couple must meet each of the following criteria:

1. The patient has received a cancer diagnosis (all malignancies will be included);
2. The patient completed cancer treatment with either curative or palliative intent ≥ 3 months earlier. Patients who currently receive hormone therapy are eligible;
3. The patient experiences severe levels of fatigue (score of ≥ 35 on the Checklist Individual Strength, subscale fatigue severity (CIS-fatigue));
4. The patient has been suffering from severe fatigue for ≥ 3 months (as self-reported by the patient);
5. The patient was ≥ 18 years old at disease onset;
6. The partner is ≥ 18 years old;
7. Both couple members live together;
8. Both couple members have good command of the Dutch language (checked implicitly during registration);
9. Both couple members have adequate computer literacy and have access to an internet-connected computer, laptop or tablet (based on self-report);
10. Both couple members agree to participate in the research.

Exclusion Criteria:

The couple will be excluded in case:

1. The patient is currently following an evidence-based therapy for CCRF (i.e. Cognitive-Behavioral Therapy, mindfulness-based therapy, exercising/physiotherapy) as self-reported at the (telephone) screening;
2. The patient suffers from a condition that can explain his/her fatigue and is potentially treatable (e.g. anemia);
3. The therapist decides, based on information collected during the intake session, that the intervention is not suitable for the couple. Criteria that will be considered include, but are not limited to:

   * presence of severe psychiatric morbidity such as suicidal ideation and/or psychosis (as assessed by the therapist at the intake session). Mild depression is not an exclusion criterion. A score of ≥ 20 on the Hospital Anxiety and Depression Scale (HADS) at T0 is considered indicative of depression. Therefore, if the patient or the partner scores ≥ 20, the therapist will determine at the intake whether the participant has suicidal ideation or suffers from other severe psychiatric morbidity. A participant (and thus the couple) will be excluded if, according to the therapist, that is the case;
   * presence of substance abuse, except for smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2024-03-21 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the couple eMBCT operationalized as intervention adherence | Throughout intervention completion, about 15-20 weeks per couple
  Operationalized as percentage of couples in which the patient completed the intervention and the partner did not drop out from it. Patients' intervention completion will be recorded in the therapist log and assessed by patient self-report. If either one satisfies the completion criterion, the couple will be considered as intervention completers.
  Benchmark: >= 60% of couples completed the intervention.
Acceptability of the couple eMBCT operationalized as satisfaction with the intervention | Throughout intervention completion, about 15-20 weeks per couple
  Quantitatively operationalized as satisfaction with the dyadic approach and the intervention overall (score >= 5 indicates satisfaction, (couples only, not therapists) as assessed at T1, 2 weeks after intervention completion.
  Benchmark: >= 70% of patients and 70% of partners indicating on the T1 questionnaire to be satisfied.
Potential efficacy on patient fatigue as assessed with the fatigue severity subscale of the Checklist Individual Strength (CIS-fatigue) from pre-intervention (T0) to 2 weeks post-intervention (T1) | From the pre-intervention baseline assessment (Timepoint 0) to the post-intervention assessment, 2 weeks after intervention completion (Timepoint 1)
  Fatigue is assessed with the Checklist Individual Strength, subscale fatigue severity (CIS-fatigue) on T0 (pre-intervention) and T1 (approx. 2 weeks after intervention completion). Eight items are rated on a 7-point scale, measuring fatigue in the preceding 2 weeks. The scale score ranges between 8 and 56, with a higher score indicating a higher level of fatigue.
  1. Change in patient fatigue. The change in fatigue from T0 to T1 is tested with a matched pairs t-test and according to the intention-to-treat principle.
     Benchmark: a statistically significant (p < .05) decrease in patient fatigue between T0 and T1.
  2. Clinically relevant change in patient fatigue. Operationalized as a reduction on the CIS-fatigue from T0 to T1 of at least 6-points.
  Benchmark: ≥ 45% of patients score on T1 at least 6 points lower than on T0.

SECONDARY OUTCOMES:
Feasibility of trial procedures operationalized as recruitment rate | Throughout study conduction, i.e. during the (planned) total of 18 months of data collection
  Benchmark:
  Recruitment rate: ≥ 3 couples included per month, averaged across both recruitment strategies.
Feasibility of trial procedures operationalized as T1 and T2 assessment adherence rate | Throughout study conduction, i.e. during the (planned) total of 18 months of data collection
  Benchmark:
  T1 and T2 adherence rate: ≥ 65% of patients and partners complete the T1 and ≥ 60% of patients and partners complete the T2 questionnaire.
Feasibility of trial procedures operationalized as diary adherence rate | Throughout study conduction, i.e. during the (planned) total of 18 months of data collection
  Diary adherence rate: ≥ 65% of diaries completed (11-14 diaries) by both patients and partners.
Potential working mechanisms of couple eMBCT | During diary period, 17-22 weeks
  Diary data will be analyzed to assess the intervention's potential working mechanisms, i.e. whether expected improvements in targeted variables co-occur with the expected reduction in patient fatigue. The putative mechanism variables are: affect, sleep, catastrophizing, partner communication, partner interactions, self-efficacy, mindfulness and closeness. Multilevel growth curve analysis will be applied to model the time slopes of the potential mechanisms and weekly fatigue over the entire diary period.
  A variable is interpreted as potential working mechanism in case the standardized covariance between the slope change factor for the outcome (fatigue) and that of the presumed mediator is significant (using a z-test where +/-1.96 is significant at the .05 level).

CONTACTS AND LOCATIONS:
Overall Officials: Mariët Hagedoorn, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - Helen Dowling Institute, Bilthoven
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes
Collected quantitative IPD (questionnaires, diaries) can potentially be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study completion and publication of outcome data.
Access Criteria: The anonymized data that support the findings of this study will become available from the principle investigators upon reasonable request, including a data analysis plan and research questions. Permission for data sharing will be asked from the medical ethical commission.

REFERENCES:
- [Derived] Muller F, van Dongen S, van Woezik R, Tibosch M, Tuinman MA, Schellekens MPJ, Laurenceau JP, van der Lee M, Hagedoorn M. A Web-Based Mindfulness-Based Cognitive Therapy for Couples Dealing With Chronic Cancer-Related Fatigue: Protocol for a Single-Arm Pilot Trial. JMIR Res Protoc. 2023 Nov 6;12:e48329. doi: 10.2196/48329. PMID 37930767
- See also: Study website (in Dutch) — http://www.hdi.nl/companion